CLINICAL TRIAL: NCT03647644
Title: Coagulation Test Changes Associated With Acute Normovolemic Hemodilution in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gregory A. Nuttall, M.D., Professor of Anesthesiology, Mayo Clinic
Other Study IDs: 16-003298
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Coagulation Disorder; Bleeding
Keywords: Cardiac Surgery; Bleeding; Transfusion; Acute Normovolemic Hemodilution
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Normovolemic Hemodilution Group: All patients enrolled in the study will undergo a perioperative cardiac surgical anesthetic care plan standardized to the current institutional protocol utilized for intraoperative medication administration. If clinically indicated and appropriate per the discretion of the anesthesiologist, Acute Normovolemic Hemodilution (ANH) blood, about 2 units, will be withdrawn from the patients and stored carefully at room temperature per standard protocol. At the conclusion of cardiopulmonary bypass and after protamine administration, Coagulation Laboratory Testing will be drawn from the patients prior to re-infusing the ANH blood and after the blood has been infused per standard institutional protocol.
  Interventions: Diagnostic Test: Coagulation Laboratory Testing
- Control Group: All patients enrolled in the study will undergo a perioperative cardiac surgical anesthetic care plan standardized to the current institutional protocol utilized for intraoperative medication administration. In this arm, ANH would be clinically appropriate, however, the anesthesiologist determined they would not have ANH preformed. At the conclusion of cardiopulmonary bypass and after protamine administration, Coagulation Laboratory Testing will be drawn from the patients and again 30 minutes later to mirror the time lapse in the ANH group.
  Interventions: Diagnostic Test: Coagulation Laboratory Testing

INTERVENTIONS:
Diagnostic Test: Coagulation Laboratory Testing — Standard coagulation testing (Platelet count, Fibrinogen, PT/INR, aPTT), and Thromboelastogram as is routine and per institutional protocol in this population.

SUMMARY:
The researchers are trying to reduce the need for blood transfusions in subjects having surgery that will involve the use of cardiopulmonary bypass. A unit of whole blood will be removed as part of their standard of care prior to going on cardiopulmonary bypass (CPB). This unit is given back to the subject post CPB. This has been shown to reduce the need for blood transfusion in patients.

DETAILED DESCRIPTION:
Subjects will be asked to allow the researchers to take the blood left over from normal standard of care blood draws and do coagulation testing. If clinically indicated, the blood, about 2 units, will be withdrawn from the subject. The researchers will also collect 8 ml (less than two teaspoons) of blood through the catheter that was placed as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a cardiac surgical procedure utilizing cardiopulmonary bypass
* Permission to use medical records in research

Exclusion Criteria:

* Unable to grant informed consent or comply with study procedure
* Patient refusal of ANH withdrawal.
* Undergoing emergency open heart-surgery
* CPB time is expected to be < 30 minutes
* Less than 18 years of age
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are those who are scheduled to undergo elective cardiac surgery. Researchers identify patients who based on our institutional practice would be candidates for ANH which has been shown to reduce bleeding and transfusion in cardiac surgical patients. These patients are consented to participate in the study, and are then followed through their operative day and laboratory results recorded. Patients are not randomized to any treatment arm as part of this study and it is up to the covering anesthesiologist as to whether or not a patient with undergo ANH or not (become a control).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Platelet count | baseline, 30 minutes after cardiopulmonary bypass
  A platelet is a tiny piece of cell that is made by breaking off of a large cell in the bone marrow. Platelets are found in the blood and spleen. They help form blood clots to slow or stop bleeding, and to help wounds heal. Also called thrombocyte. Normal platelet count ranges from 150,000 to 450,000 platelets per microliter of blood. Units: 10(9)/L
Change in Fibrinogen | baseline, 30 minutes after cardiopulmonary bypass
  Component of blood that aids in coagulation. Also known as a blood coagulation factor. Normal reference range 200-393 mg/dL.
Change in Prothrombin Time/international normalized ratio (PT/INR) | baseline, 30 minutes after cardiopulmonary bypass
  Laboratory test that measures the clotting ability of blood and is a marker for the amount and functionality of the clotting factors in the blood. Normal reference range 0.9-1.1 seconds
Change in aPTT | baseline, 30 minutes after cardiopulmonary bypass
  Laboratory test that measures the clotting ability of blood and is a marker for the amount and functionality of the clotting factors in the blood. Normal reference range 25-37 seconds.
Change in Thromboelastogram | baseline, 30 minutes after cardiopulmonary bypass
  Laboratory test that looks at the bloods ability to form a clot and the the strength of the blood clot. It looks at all the components that allow blood to clot as a whole. The visual shape of the test along with objective data provide diagnostic information about normal or abnormal conditions of blood coagulation.

SECONDARY OUTCOMES:
Allogenic Blood Transfusion | 24 hours postoperative
  The amount of Allogenic Blood Transfusion volume required as measured by number of transfused units of red blood cells, platelets, fresh frozen plasma, and cryoprecipitate.
Chest Tube Output | 24 hours postoperative
  A marker of bleeding in cardiac surgery patients is chest tube output. The amount of fluid as measured in mL's of blood accumulated in the chest tube collection device in 24 hours.
Re-operation | 24 hours postoperative
  A marker of bleeding in cardiac surgery patients is re-operation. The number of subjects who have re-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nuttall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No